CLINICAL TRIAL: NCT05290597
Title: A Phase 1, Open-label, Multicenter, Dose Escalation Study of IBI363 (PD1-IL2m) in Subjects with Advanced Solid Malignancies or Lymphomas
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Collaborators: Fortvita Biologics (USA)Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI363A101
Record Dates: First submitted 2022-01-09; First posted 2022-03-22 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Solid Malignancies or Lymphomas
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- IBI363 (Experimental): Single arm
  Interventions: Biological: IBI363

INTERVENTIONS:
Biological: IBI363 — a mutated IL-2 cytokine fused to an anti-PD-1 antibody to combine IL-2 pathway stimulation with checkpoint blockade.

SUMMARY:
This is a Phase 1, open-label, multicenter, dose-escalation study designed to evaluate the safety, tolerability, and DLTs to establish the maximum tolerated dose (MTD) or maximum administered dose (MAD), and the RP2D of sequential doses of IBI363 (study drug) in subjects with advanced, refractory solid malignancies or lymphomas.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, ≥ 18 years
2. Subjects with a documented (histologically- or cytologically-proven) solid tumor malignancy that is locally advanced or metastatic; subjects with documented lymphomas
3. Subjects with a malignancy (solid tumor or lymphoma) that is currently not amenable to surgical intervention due to either medical contraindications or non-resectability of the tumor
4. Subjects who are refractory to or intolerant to existing therapy(ies) known to provide clinical benefit Note: Subjects may have received and failed prior therapy with a PD-1/PD-L1 inhibitor and be considered eligible for this trial.
5. Subjects with measurable or non-measurable disease according to RECIST v1.1 or standard criteria for lymphoma (Lugano 2014)
6. Subjects, both male and female, who are either not of childbearing potential or who agree to use a highly effective method of contraception during the study beginning within 2 weeks prior to the first dose and continuing until 6 months after the last dose of study drug
7. Subjects with the ability to understand and give written informed consent for participation in this trial, including all evaluations and procedures as specified by this protocol

Exclusion Criteria:

1. Women who are pregnant or lactating, or intending to become pregnant before, during, or within 6 months after the last dose of study drug. Women of childbearing potential (WOCBP) or fertile men with WOCBP partner(s), not using and not willing to use a highly effective method of contraception.
2. Subjects with history of or known active seizure disorder, brain metastases, spinal cord compression, or carcinomatous meningitis, or new evidence of brain or leptomeningeal disease.
3. Subjects with:

   * Active thrombosis, or a history of deep vein thrombosis (DVT) or pulmonary embolism (PE) within 4 weeks prior to first administration of study drug unless adequately treated and considered by the Investigator to be stable.
   * Active uncontrolled bleeding or a known bleeding diathesis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of serious adverse events (SAEs), treatment-emergent AEs (TEAEs) and immune-related AEs (irAEs) | up to 90 days after the last administration
  An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly/birth defect or is an important medical event that may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed before. A TEAE will be defined as any new AE that begins, or any pre-existing condition that worsens in severity, after at least 1 dose of study treatment has been administered. irAEs will be assessed.
Number of participants with abnormality in vital signs | up to 90 days after the last administration
  Blood pressure, pulse, respiratory rate, and temperature will be assessed.
Number of participants with abnormality in hematology parameters | up to 90 days after the last administration
  Blood samples will be collected to evaluate hemoglobin, mean corpuscular volume (MCV), white blood cell (WBC) count, platelets, 5-part differential white cell count, mean platelet volume and coagulation factors including international normalized ratio (INR), activated partial thromboplastin time (aPTT) and prothrombin time (PT)
Number of participants with abnormality in clinical chemistry parameters | up to 90 days after the last administration
  Blood samples will be collected to evaluate sodium, potassium, calcium, magnesium, chloride, glucose, creatinine, urea or blood urea nitrogen (BUN), bicarbonate, amylase, bilirubin, alkaline phosphatase, aspartate aminotransferase (AST), alanine aminotransferase (ALT), total protein, albumin, lactate dehydrogenase and lipase.
Number of participants with abnormality in routine urinalysis parameters | up to 90 days after the last administration
  Urine samples will be collected to evaluate specific gravity, leucocyte esterase, nitrite, blood, bilirubin, protein, glucose, ketones and urobilinogen.
Number of participants with abnormality in ECG parameters | up to 90 days after the last administration
  12-lead ECG will be obtained using an ECG machine. Participants will be in supine or a semi-recumbent position (about 30 degrees of elevation) and rested for approximately 2 minutes before ECGs are recorded.
Number of dose-limiting toxicity (DLT) | 28 days during the first 4-week cycle
  Incidence of dose-limiting toxicity (DLT) events

SECONDARY OUTCOMES:
maximum concentration (Cmax) | Up to 2 years
  PK parameters to be evaluated for IBI363 including maximum concentration (Cmax) will be determined when appropriate.
area under the curve (AUC) | Up to 2 years
  PK parameters to be evaluated for IBI363 including area under the curve (AUC) will be determined when appropriate.
clearance (CL) | Up to 2 years
  PK parameters to be evaluated for IBI363 including area under the curve (AUC) will be determined when appropriate.
half-life (t1/2) of IBI363 | Up to 2 years
  PK parameters to be evaluated for IBI363 including volume of distribution (V) will be determined when appropriate.
Objective response rate (ORR) | Up to 2 years
  To evaluate the preliminary antitumor activity of IBI363
time to response (TTR) | Up to 2 years
  To evaluate the preliminary antitumor activity of IBI363
duration of response (DoR) | Up to 2 years
  To evaluate the preliminary antitumor activity of IBI363
disease control rate (DCR) | Up to 2 years
  To evaluate the preliminary antitumor activity of IBI363
progression-free survival (PFS) | Up to 2 years
  To evaluate the preliminary antitumor activity of IBI363
6-month and 1-year PFS rate per RECIST v1.1 for subjects with solid tumors, and per Lugano 2014 for subjects with lymphomas | Up to 2 years
  To evaluate the preliminary antitumor activity of IBI363
Overall survival (OS) | through study completion, an average of 1 year
  To evaluate the preliminary antitumor activity of IBI363
survival rates (6-month and 1-year) | Up to 2 years
  To evaluate the preliminary antitumor activity of IBI363
The incidence of ADA and NAb of IBI363 | Up to 2 years
  Each subject will be tested for anti-drug (IBI363) antibody (ADA), and ADA-positive serum samples will continue to be tested for neutralizing antibodies (NAb).

CONTACTS AND LOCATIONS:
Overall Officials: Morteza Aghmesheh, Principal Investigator — Southern Medical Day Care Centre
Locations (4):
- Australia (4):
  - Kate.Wilkinson1@health.nsw.gov.au, Sydney, New South Wales
  - Westmead Hospital, Sydney, New South Wales
  - Sydney Southwest Private Hospital, Sydney, New South Wales
  - Cancer Care Wollongong, Sydney, New South Wales

IPD SHARING:
Plan to Share IPD: No